CLINICAL TRIAL: NCT01277328
Title: Tocilizumab (RoActemra) poST Marketing Observational Study in DMARD-IR Patients to Assess Efficacy and Safety in routiNE Clinical Practice - STONE
Brief Title: An Observational Study of RoActemra/Actemra (Tocilizumab) in Patients With Rheumatoid Arthritis
Status: Terminated | Type: Observational
Why Stopped: Contract terminated with Site Management Organization
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25332
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort: Cohort

SUMMARY:
This observational, prospective, open-label, multi-center study will evaluate the effectiveness in disease reduction and the safety of RoActemra/Actemra (tocilizumab) in patients with rheumatoid arthritis. Data will be collected for 11 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >/=18 years of age
* Patients with rheumatoid arthritis eligible for RoActemra

Exclusion Criteria:

* Hypersensitivity to RoActemra
* Active, severe infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis receiving RoActemra/Actemra
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Mean change in Disease Activity Score 28 (DAS28) | 11 months

SECONDARY OUTCOMES:
Proportion of patients with a change in Disease Activity Score 28 (DAS28) | 5 months
European League Against Rheumatism (EULAR) response rates | 20 weeks
Proportion of patients with disease remission | 20 weeks
Proportion of patients with low disease activity | 20 weeks
Incidence of adverse events | 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Bucharest, Romania